## NCT07211698

# A QUALITATIVE STUDY EXPLORING ETHNIC MINORITIES' EXPERIENCES OF HEALTHCARE INTERVENTIONS DELIVERED AT HOME OR IN COMMUNITY CENTRES

Ethnic Minorities' Experiences of Healthcare Intervention

27 OCTOBER 2025





## **INFORMED CONSENT FORM (WRITTEN)**

Version 3.0, 27.10.2025 REC ref: FMHS 212-0725

Participant number: \_\_\_\_\_

Chief Investigator: Dr Katie Robinson

Please write your initials on the box to confirm.

| information | | 1 |
|---|---|---|
| 1. | I have <b>read and understand</b> the <b>information</b> sheet <i>PIS version 3.0</i> dated 27.10.2025 for the above study and I confirm I have had the opportunity to ask questions. | |
| volunteering | | |
| <b>1</b> 2. | I <b>understand</b> that <b>taking part</b> is my <b>choice</b> and that I am <b>free to withdraw</b> at <b>any time</b> . | |
| stop<br>3. | I understand that if I withdraw, any information collected about me up until this point will be kept and used in the final study report. | |
| checking | | |
| 4. | I understand that the results of the interview may be looked by someone not part of the study team to check that the study is being carried out correctly as required by UK law. | |
| torgerint torgerint torgering to the second | I consent to the use of an interpreter, direct quotes, fieldnotes, audio recording, and transcription of the interview. | |



| contact information kept safe kept safe | I <b>consent</b> to the <b>storage</b> of my <b>personal information</b> for the purposes of this study including on a computer. |
|---|---|
| 7. | I <b>understand</b> that any <b>information</b> that could identify me will be <b>kept confidential</b> and no personal information will be included in the study report or other publications. |
| do not share information 8. | I <b>agree not to disclose</b> anything that has been discussed during the study <b>conversations outside</b> of the <b>study</b> . |
| agree | I <b>agree</b> to <b>take part</b> in the <b>study</b> . |
| /・ | |
| | Optional |
| private information 10. | Optional I am happy for the researcher to have my contact information to get in touch with what the study found. |
| | I am happy for the researcher to have my contact information to get in touch with what the study |



# Participants contact details

| Telephone: | | |
|---|---|---|
| Email: | | |
| Postcode NOT your full address: | | |
| Name of participant: | Participant's signature: | Date: |
| First Name and Surname<br>(BLOCK CAPITALS) | | |
| Name of researcher: | Researcher's signature: | Date: |
| First Name and Surname<br>(BLOCK CAPITALS) | | |



### FOR WITNESS OR INTERPRETER/TRANSLATOR USE ONLY

Complete this section if participant is not able to read the study information and/or sign for themselves but has capacity to give consent OR if the study information has been interpreted or translated to the participant.

| WITNESS STATEMENT: | | |
|---|---|---|
| I witnessed accurate reading of the consent form to the potential participant, who could ask any questions and received satisfactory answers | | |
| I confirm that participant gave their consent freely. | | |
| Witness First Name and Surname (BLOCK CAPITALS) | Signature | Date |

### INTERPRETER/TRANSLATOR STATEMENT:

I was present during the meeting between the researcher Joy Watterson and the participant. I translated/interpreted information for the participant.

I confirm that study information was interpreted/translated accurately.

| Interpreter/translator | Signature | Date |
|--------------------------------------------|-----------|------|
| First Name and Surname<br>(BLOCK CAPITALS) | | |